CLINICAL TRIAL: NCT07221656
Title: Evaluation of Prolonged Asparaginase Activity Levels After Calaspargase Pegol Administration
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-009034; NCI-2025-07667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-009034 (Other: Mayo Clinic)
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients provide blood samples collected during regularly scheduled appointments and have medical records reviewed throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates the median duration of therapeutic serum asparaginase activity (SAA) levels after administration of calaspargase pegol (Cal-PEG) and the potential association between peak SAA levels and duration of therapeutic levels with toxicity in pediatric patients with acute lymphoblastic leukemia or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia/lymphoma being treated by the pediatric hematology team
* Receiving calaspargase as part of treatment for malignancy

Exclusion Criteria:

* Age > 21 years
* Patients who are actively enrolled on Children's Oncology Group (COG) trial AALL1732 in an inotuzumab containing arm
* Pregnancy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute lymphoblastic leukemia/lymphoma being treated by the pediatric hematology team at Mayo Clinic in Rochester
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of therapeutic SAA | Up to 15 months
  Descriptive statistics including medians and interquartile ranges will be utilized to summarize continuous variables.

OTHER OUTCOMES:
Asparaginase-related toxicities correlated with duration of therapeutic SAA levels | Up to 15 months
  Spline plots will be used to assess any correlation between duration of therapeutic SAA levels and incidence of asparaginase-associated toxicities. Categorical data including toxicity information will be summarized descriptively. Toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, per standard of care.
Asparaginase-related toxicities correlated with peak SAA levels | Up to 15 months
  Spline plots will be used to assess any correlation between peak SAA levels and incidence of asparaginase-associated toxicities. Categorical data including toxicity information will be summarized descriptively. Toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, per standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine B. O'Keefe, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials